CLINICAL TRIAL: NCT00000187
Title: Ritanserin in Treatment of Cocaine Dependence
Brief Title: Ritanserin in Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, James Cornish, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-00144-1; 3R01DA012268 (NIH); K20-00144-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Dependence; ritanserin
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ritanserin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Ritanserin

SUMMARY:
The purpose of this study is to assess ritanserin as a pharmacotherapy for cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Ages: 28 Years to 47 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 1992-07; Primary Completion 1994-06 (Actual)

PRIMARY OUTCOMES:
Cocaine use
Cocaine craving

CONTACTS AND LOCATIONS:
Overall Officials: James Cornish, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cornish JW, Maany I, Fudala PJ, Ehrman RN, Robbins SJ, O'Brien CP. A randomized, double-blind, placebo-controlled study of ritanserin pharmacotherapy for cocaine dependence. Drug Alcohol Depend. 2001 Jan 1;61(2):183-9. doi: 10.1016/s0376-8716(00)00140-x. PMID 11137283